CLINICAL TRIAL: NCT06911073
Title: A Double-Blind, Randomized Placebo-Controlled Study to Evaluate a Postbiotic Supplement in Supporting Weight Loss and Metabolic Health
Brief Title: A Study to Evaluate a Postbiotic in Supporting Weight Loss and Metabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ResBiotic Nutrition, Inc. (Industry)
Collaborators: Able Biolabs, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ABL-032501
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Obesity and Overweight
Keywords: Postbiotic; Obesity; GLP-1; Metabolic health
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Randomization at 1:1 ratio of active:placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 1 capsule of placebo, taken once daily
  Interventions: Dietary Supplement: Placebo
- Postbiotic Supplement (Experimental): 1 capsule of 40 mg postbiotic, 450 mg herbal blend, and 810 mcg vitamins taken once daily
  Interventions: Dietary Supplement: Postbiotic

INTERVENTIONS:
Dietary Supplement: Postbiotic — Active ingredients:
  Vitamin D (as cholecalciferol) - 10 mcg Vitamin B12 (as methylcobalamin) - 200 mcg Chromium (as chromium picolinate) - 600 mcg resM™ Postbiotic (L. plantarum RSB11® HI - 16B cells) - 40 mg White mulberry (Morus alba) leaf extract - 250 mg Fenugreek (Trigonella foenum-graecum) seed extract - 200 mg
  Inactive ingredients:
  Microcrystalline cellulose, hydroxypropyl methylcellulose, magnesium stearate, silica, water, carrageenan, potassium acetate
  Other Names: resM™ GLP-1 Postbiotic
  Arms: Postbiotic Supplement
Dietary Supplement: Placebo — Active ingredients:
  N/A
  Inactive ingredients:
  Microcrystalline cellulose, hydroxypropyl methylcellulose, magnesium stearate, silica, water, carrageenan, potassium acetate
  Arms: Placebo

SUMMARY:
This study aims to evaluate the impact of a specific oral postbiotic supplement on metabolic health in overweight adults.

DETAILED DESCRIPTION:
Obesity poses substantial health challenges contributing significantly to chronic metabolic disorders such as type 2 diabetes mellitus, cardiovascular disease, and diminished quality of life for people worldwide. Central to obesity-related metabolic dysfunction is dysregulation of appetite control, glucose homeostasis, insulin sensitivity, and systemic inflammation. Evidence indicates a strong connection between these metabolic disturbances and alterations in the gut microbiome, implicating microbiota dysbiosis as a potential target for intervention. Microbiome-based interventions underscore a promising approach in weight management and metabolic health.

ELIGIBILITY:
Inclusion Criteria:

1. Provide voluntary signed and dated informed consent.
2. Be in good health as determined by medical history.
3. Age between 18 and 65 yr (inclusive).
4. Body Mass Index of 25.0 - 40.0 (inclusive).
5. Subject agrees to maintain existing dietary and physical activity patterns throughout the study period.
6. Agree to refrain from other probiotic and postbiotic supplement products throughout the duration of the trial.
7. Subject is willing and able to comply with the study protocol.
8. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

1. History of unstable or new-onset cardiovascular/cardiorespiratory, liver, or renal conditions.
2. Alcohol abuse (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) or drug abuse or dependence within the past 6 months.
3. Previous bariatric surgery.
4. Current smokers or smoking within the past month.
5. History of hyperparathyroidism or an untreated thyroid condition.
6. History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
7. Other known gastrointestinal or metabolic conditions that might impact nutrient absorption or metabolism, e.g., short bowel syndrome, irritable bowel syndrome (IBS), diarrheal illnesses, history of colon resection, gastroparesis, Inborn-Errors-of-Metabolism (such as PKU).
8. Chronic inflammatory condition (e.g., rheumatoid arthritis, Crohn's, ulcerative colitis, Lupus, HIV/AIDS, etc.).
9. Previous medical diagnosis of gout or fibromyalgia.
10. Pregnant women, women trying to become pregnant, women less than 120 days postpartum or nursing women. Any woman that is sexually active will have to take report their pregnancy status prior to enrolling and during the trial if they become pregnant.
11. Known sensitivity to any ingredient in the test formulations as listed in the product label.
12. Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of resM™ on weight | 8 weeks
  Change from baseline in weight (lb)
To determine the effect of resM™ on BMI | 8 weeks
  Change from baseline in BMI. Weight and height will be combined to report BMI in kg/m^2)
To determine the effect of resM™ on food cravings | 8 weeks
  Change in reported food cravings from baseline based on Food Craving Questionnaire Trait-reduced (FCQ-T-r) scores. The total score reflects the severity of food cravings where 90 indicates the most severe and 15 indicates the least severe.
To determine the effect of resM™ on blood metabolic markers | 8 weeks
  Change from baseline in serum fasting glucose
To determine the effect of resM™ on blood metabolic markers | 8 weeks
  Change from baseline in serum insulin levels
To determine the effect of resM™ on blood metabolic markers | 8 weeks
  Change from baseline in whole blood HbA1c (glycated hemoglobin)

SECONDARY OUTCOMES:
To determine the effect of resM™ on GLP-1 | 8 weeks
  Change from baseline in plasma active and inactive GLP-1 protein
To determine the effect of resM™ on DPP-4 | 8 weeks
  Change from baseline in plasma DPP4
To determine the effect of resM™ on gut microbiome | 8 weeks
  Change from baseline in gut microbiome as assessed by 16s metagenomic sequencing on fecal samples
To determine the effect of resM™ on depression | 8 weeks
  Change from baseline in reported depression levels based on Patient Health Questionnaire 9 (PHQ-9) scores. The total score reflects the severity of depression where 1 indicates minimal depression and 27 indicates severe depression.
Change in Albumin after taking resM™ | 8 weeks
  Change from baseline in Albumin
Change in Albumin/Globulin ratio after taking resM™ | 8 weeks
  Change from baseline in Albumin/Globulin ratio
Change in Alkaline Phosphatase after taking resM™ | 8 weeks
  Change from baseline in Alkaline Phosphatase
Change in Alanine Aminotransferase (ALT) after taking resM™ | 8 weeks
  Change from baseline in Alanine Aminotransferase (ALT)
Change in Aspartate Aminotransferase (AST) after taking resM™ | 8 weeks
  Change from baseline in Aspartate Aminotransferase (AST)
Change in BUN/Creatinine ratio after taking resM™ | 8 weeks
  Change from baseline in blood urea nitrogen (BUN)/creatinine ratio
Change in Calcium after taking resM™ | 8 weeks
  Change from baseline in calcium
Change in Chloride after taking resM™ | 8 weeks
  Change from baseline in chloride
Change in Glucose after taking resM™ | 8 weeks
  Change from baseline in glucose
Change in Sodium after taking resM™ | 8 weeks
  Change from baseline in sodium
Change in Total Bilirubin after taking resM™ | 8 weeks
  Change from baseline in total bilirubin
Change in Total Protein after taking resM™ | 8 weeks
  Change from baseline in total protein
Change in Urea Nitrogen after taking resM™ | 8 weeks
  Change from baseline in Urea Nitrogen
Change in White Blood Cell (WBC) count after taking resM™ | 8 weeks
  Change from baseline in white blood cell (WBC) count
Change in Red Blood Cell (RBC) count after taking resM™ | 8 weeks
  Change from baseline in red blood cell (RBC) count
Change in Hemoglobin (Hb) after taking resM™ | 8 weeks
  Change from baseline in hemoglobin (Hb)
Change in Hematocrit (Hct) after taking resM™ | 8 weeks
  Change from baseline in hematocrit (Hct)
Change in Mean Corpuscular Volume (MCV) after taking resM™ | 8 weeks
  Change from baseline in mean corpuscular volume (MCV)
Change in Mean Corpuscular Hemoglobin (MCH) after taking resM™ | 8 weeks
  Change from baseline in mean corpuscular hemoglobin (MCH)
Change in Mean Corpuscular Hemoglobin Concentration (MCHC) after taking resM™ | 8 weeks
  Change from baseline in mean corpuscular hemoglobin concentration (MCHC)
Change in Red Cell Distribution Width (RDW) after taking resM™ | 8 weeks
  Change from baseline in red cell distribution width (RDW)
Change in Platelet Count after taking resM™ | 8 weeks
  Change from baseline in platelet count
Change in Mean Platelet Volume (MPV) after taking resM™ | 8 weeks
  Change from baseline in Mean Platelet Volume (MPV)
Change in Neutrophils after taking resM™ | 8 weeks
  Change from baseline in neutrophil count (absolute) and differential (percent)
Change in Lymphocytes after taking resM™ | 8 weeks
  Change from baseline in lymphocyte count (absolute) and differential (percent)
Change in Monocytes after taking resM™ | 8 weeks
  Change from baseline in monocyte count (absolute) and differential (percent)
Change in Eosinophils after taking resM™ | 8 weeks
  Change from baseline in eosinophil count (absolute) and differential (percent)
Change in Basophils after taking resM™ | 8 weeks
  Change from baseline in basophil count (absolute) and differential (percent)
Safety - participants experiencing adverse events | 8 weeks
  The number of participants experiencing Treatment Emergent Adverse Events (TEAEs)
Safety - total adverse events | 8 weeks
  The total number of Treatment Emergent Adverse Events (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelgawad, MD, Principal Investigator — Able Biolabs, LLC
Locations (1):
- Able Biolabs, LLC, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No